CLINICAL TRIAL: NCT01603667
Title: PG2 Injection 500 mg in Acute Stroke Study (Pass): A Randomized, Double-Blind, Placebo-Controlled Study of PG2 Injection 500 mg in Patients With Treatment Started Within 3-6 Hrs of the Onset of Acute Ischemic Stroke
Brief Title: PG2 Injection 500 mg in Acute Stroke Study (Pass)
Acronym: Pass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); Tri-Service General Hospital (Other); Changhua Christian Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University (Other); En Chu Kong Hospital (Other); Kuang Tien General Hospital (Other); Chung Shan Medical University (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Kaohsiung Veterans General Hospital. (Other); Taipei Medical University Shuang Ho Hospital (Other); Cheng Hsin Rehabilitation Medical Center (Other); Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMR100-IRB-185
Record Dates: First submitted 2012-05-20; First posted 2012-05-22 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PG2 Injection 500 mg (Experimental): PG2 Injection 500 mg
  Interventions: Drug: PG2
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PG2 — STUDY DRUG DOSAGE:IV infusion of PG2 Injection 500 mg in 500 ml Normal Saline at a rate of 200 mg/hr with infusion started within 3-6 hrs of stroke onset and infusion of a total of 500 mg PG2 Injection in 500 ml Normal Saline or 500 ml Normal Saline will be completed within 2.5~3.5 hrs. The same dose of PG2 Injection 500 mg will be repeated daily for the subsequent 2 days.
  ROUTE OF ADMINISTRATION:Continuous IV infusion via a calibrated infusion pump DURATION FOR EACH PATIENT:90 days
  Other Names: Polysaccharides of Astragalus membranaceus
  Arms: PG2 Injection 500 mg
Drug: placebo — STUDY DRUG DOSAGE: IV infusion of Placebo Injection 500 mg in 500 ml Normal Saline at a rate of 200 mg/hr with infusion started within 3-6 hrs of stroke onset and infusion of a total of 500 mg Placebo Injection in 500 ml Normal Saline or 500 ml Normal Saline will be completed within 2.5~3.5 hrs. The same dose of Placebo Injection 500 mg will be repeated daily for the subsequent 2 days.
  ROUTE OF ADMINISTRATION:Continuous IV infusion via a calibrated infusion pump DURATION FOR EACH PATIENT:90 days
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of PG2 Injection 500 mg versus placebo, administered intravenously within 3-6 hrs of stroke onset to patients with an acute ischemic stroke, as determined by Modified Rankin Scale (mRS) score at Day 90.

The secondary objectives are as follows:

* To evaluate the efficacy of PG2 Injection 500 mg versus placebo as determined by Barthel Index (BI) score at Day 90.
* To evaluate the efficacy of PG2 Injection 500 mg in reducing the risk of recurrent stroke, cardiovascular events and death of all causes.
* To evaluate the safety of PG2 Injection 500 mg treatment

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled multi-center study of intravenous (IV) PG2 Injection 500 mg starting within 3-6 hrs of the onset of acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with acute ischaemic stroke
2. Patient, or a family member with legally authorized responsibility, has given informed consent
3. Age ≥20 years
4. Infusion of study medication can be started within 3-6 hrs of stroke onset.
5. NIHSS score of ≥ 7 - 24

Exclusion Criteria:

1. Intracranial haemorrhage (ICH) identified by CT or MRI
2. Rapidly improving symptoms, particularly if in the judgment of the managing clinician that the improvement is likely to result in the patient having an NIHSS score of < 6 at randomization
3. Pre-stroke mRS score of ≥ 2 (indicating previous disability)
4. Known allergy to Astragalus membranaceus or its mayor derivatives (polysaccharides)
5. Patients who are eligible for tPA treatment and has been treated with tPA.
6. Participation in any investigational study in the previous 30 days
7. Any terminal illness such that patient would not be expected to survive more than 1 year
8. Any condition that could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study (this applies to patients with severe microangiopathy such as haemolytic uremic syndrome or thrombotic thrombocytopenic purpura). The judgment is left to the discretion of the Investigator
9. Pregnant women (clinically evident)
10. Previous stroke within last three months
11. Past history or clinical presentation of ICH, arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm.
12. Current use of oral anticoagulants with prolonged prothrombin time (INR > 1.6)
13. Use of heparin, except for low dose subcutaneous heparin, in the previous 48 hrs and a prolonged activated partial thromboplastin time exceeding the upper limit of the local laboratory normal range
14. Clinically significant hypoglycaemia (blood sugar < 50mg/dl)
15. Uncontrolled hypertension defined by a blood pressure > 185 mmHg systolic or >110 mmHg diastolic on at least 2 separate occasions at least 10 minutes apart, or requiring aggressive treatment to reduce the blood pressure to within these limits. The definition of "aggressive treatment" is left to the discretion of the responsible Investigator
16. Major surgery within the preceding 14 days which poses risk in the opinion of the Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the percentage of patients who are categorized as good functional outcome with mRS <2 | 90 days

SECONDARY OUTCOMES:
Percentage of patients who achieve a Day 90 BI score of 95-100 Percentage of patients who are free of recurrent stroke, cardiovascular events and death of all causes. Percentage of patients who are free of adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Chung Y. Hsu, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan